CLINICAL TRIAL: NCT02958904
Title: Association Between Depressive Symptoms and Sexual Dysfunction in Men With Traumatic Spinal Cord Injury
Brief Title: Depressive Symptoms and Sexual Dysfunction in Traumatic Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Josepha Karinne de Oliveira Ferro, Master degree, Universidade Federal de Pernambuco
Other Study IDs: Depressive symptoms SCI
Record Dates: First submitted 2016-11-06; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Cord Injuries; Male Sexual Dysfunction
Keywords: Sexuality; Spinal cord injuries; Erectile dysfunction; depression
MeSH Terms: conditions — Spinal Cord Injuries; Sexuality; Erectile Dysfunction; Depression

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: using questionnaires — using questionnaires International Index Erectile Function and Beck Depression Inventory.

SUMMARY:
Aims: assess the relationship between sexual function and depressive symptoms in individuals with spinal cord injury.

DETAILED DESCRIPTION:
Method: Observational study of 44 men with spinal cord injury, age above 18 years, injury time more than six months, sexually active and accompanied in Recife referral hospitals. The degree of neurological impairment was assessed using the revised version in 2011 ASIA Impairment Scale (AIS), depressive symptoms were detected by the Beck Depression Inventory, and the evaluation of sexual function was obtained through the Erectile Function of International Index (IIEF). Descriptive statistics and bivariate analysis to assess the association were applied, with 0,05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of traumatic spinal cord injury
* injury time less than six months
* sexually active

Exclusion Criteria:

* patients who had erectile dysfunction attributed to endocrine or metabolic disease order
* those who underwent surgery in the genital area, such as radical prostatectomy or penile implant
* cognitive impairment

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included 44 men, aged between 18 and 60 years with a clinical diagnosis of traumatic spinal cord injury, injury time less than six months heterosexual and sexually active. The study excluded patients who had erectile dysfunction attributed to endocrine or metabolic disease order, those who underwent surgery in the genital area, such as radical prostatectomy or penile implant and cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
depressive symptoms | one day
  Depressive symptoms assessed by Beck Depression Inventory (BDI)

SECONDARY OUTCOMES:
Level of neurological lesion | one day
  Level of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Degree of neurological lesion | one day
  Degree of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Male Sexual Dysfunction | one day
  Male Sexual Dysfunction assessed by International Index of Erectile Function (IIEF)

IPD SHARING:
Plan to Share IPD: No